CLINICAL TRIAL: NCT04014296
Title: Effects of Dietary Protein Intake and Resistance Training on Retention of Fat Free Mass During Weight Loss in Adults Over 50 with Obesity
Brief Title: Weight Loss in Adults Over 50 with Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Drew Sayer, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB-300003818
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: weight loss; dietary protein; exercise training; fat free mass
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet, High-Protein; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Protein Diet (Experimental): Enrollment in State of Slim (SOS) weight loss program with a high protein diet.
  Interventions: Behavioral: High Protein Diet
- Resistance Training (Experimental): Enrollment in State of Slim (SOS) weight loss program with resistance training counseling sessions.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: High Protein Diet — 16 week group-based weight loss program with high protein diet. Approximate macronutrient distributions (carbohydrate:protein:fat) will be 32%:40%:28%. Because this protocol uses a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed after 8 weeks. Non-responders will be randomized to either combine the HP diet with supervised resistance training counseling (2 days per week) or add a protein supplement.
  Arms: High Protein Diet
Behavioral: Resistance Training — 16 week weight loss program with normal protein diet and resistance training counseling. Approximate macronutrient distributions (carbohydrate:protein:fat) will be 53%:20%:26%. Because this protocol uses a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed after 8 weeks. Non-responders will be randomized to either combine resistance training with HP/protein supplement or add supervised sessions with a personal trainer (2 days per week) to the resistance training regimen.
  Arms: Resistance Training

SUMMARY:
The purpose of this study is to examine the separate and combined effects of a high-protein (HP) diet and resistance training (RT) on body composition and potential biological moderators of body weight in women and men >50y. All participants will receive dietary physical activity guidance through our group-based weight loss program, State of Slim (SOS). The SOS program will be delivered via the Zoom videoconferencing platform. These participants will be randomized to receive either a counseling-based HP diet plan or RT plan. Body composition assessments at 8 wk will identify responders and non-responders; the latter will be re-randomized to "augment" (HP: add protein supplements; RT: supervise RT) or "combine" (HP with protein supplements + supervised RT).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥50 years
* Post-menopausal if Female
* BMI of 30-50 kg/m2 for ambulatory participants (less than or equal to 350 lbs.)
* BMI of 25-50 kg/m2 for wheelchair users (less than or equal to 350 lbs.)
* Ambulatory with or without a walking device or use of a manual wheelchair for mobility.

Exclusion Criteria:

* Untreated hyper or hypothyroidism.
* Cancer (except basal cell).
* Gastrointestinal disorders affecting food intake.
* <3 months of stable use of medications that affect metabolism, body weight, energy expenditure or appetite.
* Current eating disorder (e.g., binge eating disorder, anorexia, or bulimia).
* Any medical condition for which following a HP diet and/or 70 minutes of exercise daily would be inadvisable.
* Uses a powered wheelchair for mobility.
* Has a pacemaker or any other life-sustaining medical implant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment and Retention Rates | Baseline through week 52.
  Rates of study recruitment and retention will be tracked to determine clinical trial feasibility.
Class Attendance | Baseline through week 52.
  Class Attendance will be tracked to determine clinical trial feasibility.
1st Stage Treatment Credibility | Baseline.
  Perceived credibility of 1st stage interventions will be measured at baseline with the Credibility/Expectancy Questionnaire.
2nd Stage Treatment Credibility | Week 8.
  Perceived credibility of 2nd stage interventions will be measured in non-responders to 1st stage interventions at week 8 with the Credibility/Expectancy Questionnaire.
1st Stage Intervention Preference | Baseline
  Participant preferences for 1st stage interventions will be measured at baseline by answering a 5-point Likert question with '1' and '5' representing a strong preference for either intervention and '3' representing no intervention preference.
2nd Stage Intervention Preference | Week 8
  Participant preferences for 2nd stage interventions will be measured at week 8 by answering a 5-point Likert question with '1' and '5' representing a strong preference for either intervention and '3' representing no intervention preference.

SECONDARY OUTCOMES:
Body Weight | Baseline, Weeks 8, 16, and 52
  Changes from baseline body weight will be measured at weeks 8, 16, and 52.
Fat mass | Baseline, Weeks 8, 16, and 52
  Changes from baseline fat mass will be measured at weeks 8, 16, and 52.
Fat free mass | Baseline, Weeks 8, 16, and 52
  Changes from baseline fat free mass will be measured at weeks 8, 16, and 52.

OTHER OUTCOMES:
Change in glucose | Baseline to Weeks 8, 16, and 52
  Serum glucose will be measured in a fasted state and after a glucose load [mg/dL]
Change in insulin | Baseline to Weeks 8, 16, and 52
  Serum insulin will be measured in a fasted state and after a glucose load, measured in micro-units/milliliter [uU/mL]
Changes in lipids | Baseline to Weeks 8, 16, and 52
  Fasting serum concentrations of total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides
Changes in disposition index | Baseline to Weeks 8, 16, and 52
  Derived from Oral Glucose Tolerance Test (OGTT) using 0 minute and 30 minute time-points.
Changes in aerobic fitness | Baseline to Weeks 8, 16, and 52
  6-Minute Walk test for ambulatory participants OR 6-Minute Push test for wheelchair users.
Changes in physical activity | Baseline to Weeks 8, 16, and 52
  7-day accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Drew Sayer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No